CLINICAL TRIAL: NCT05846880
Title: EVALUATION OF CHOLECALCIFEROL (VitD3) MAINTENANCE SUPPLEMENTATION IN PATIENTS WITH MULTIPLE MYELOMA (MM) UNDERGOING TRANSPLANTATION AND IN COMBINATION WITH LENALIDOMIDE MAINTENANCE
Brief Title: VitD3 Supplementation in Patients With Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Amany Keruakous, MD, MS. (Other)
Responsible Party: Sponsor-Investigator, Amany Keruakous, MD, MS., Assistant Professor of Medicine, Augusta University
Organization: Augusta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCC-22-044
Record Dates: First submitted 2023-02-08; First posted 2023-05-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Myeloma, Multiple; Vitamin D; Vitamins; Lenalidomide; Revlimid; Cholecalciferol; Transplantation, Autologous; Vitamin D Deficiency
MeSH Terms: conditions — Multiple Myeloma; Vitamin D Deficiency | interventions — Lenalidomide; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance Vitamin D (Experimental): In this arm, patients will receive maintenance Vitamin D3 prior to autologous transplantation (ASCT). Within 120 days after ASCT the following will be assessed: vitamin D level, Overall Response Rate (ORR) and Measurable Residual Disease (MRD). Then patients will receive lenalidomide and continuation of maintenance Vitamin D.
  Interventions: Drug: Lenalidomide; Drug: Maintenance Vitamin D
- No Maintenance Vitamin D (Active Comparator): In this arm, patients will receive no maintenance vitamin D prior to ASCT. Within 120 days after ASCT the following will be assessed: vitamin D level, ORR, and MRD. Then patients will receive the standard lenalidomide dose along with no maintenance vitamin D.
  Interventions: Drug: Lenalidomide; Drug: No maintenance Vitamin D

INTERVENTIONS:
Drug: Lenalidomide — For first three cycles, taken orally once daily for 28 days at 10mg/day dose. After cycle 4, taken orally once daily at 15 mg/day dose
  Other Names: Revlimid
Drug: Maintenance Vitamin D — After replacement of vitamin D deficiency with weekly cholecalcefirol 50,000 units untill levels are > 30, will start maintenance therapy with Monthly replacement with 50,000 IU
  Other Names: Cholecalciferol
  Arms: Maintenance Vitamin D
Drug: No maintenance Vitamin D — After replacement of vitamin D deficiency with weekly cholecalcefirol 50,000 units untill levels are > 30, stop replacement and continue monitoring levels
  Other Names: Cholecalciferol
  Arms: No Maintenance Vitamin D

SUMMARY:
The goal of this clinical trial is to evaluate post-transplant immune reconstitution and lymphocyte recovery as well as the 3-year progression-free survival of patients with multiple myeloma in two treatment arms. One arm will receive Maintenance Vitamin D and the other arm will receive no maintenance Vitamin D prior to ASCT. Post ASCT arm 1 will have lenalidomide and maintenance VitD, and arm 2 will receive lenalidomide and no maintenance VitD. This clinical trial will also evaluate the overall response rate and survival for both treatment arms.

DETAILED DESCRIPTION:
Management of multiple myeloma (MM) has changed significantly over the past 10 years. The use of three drug induction therapy followed by autologous stem cell transplantation (ASCT) has become standard of care for transplant eligible patients with MM since randomized trials showed improved progression-free survival (PFS) and overall survival (OS) with three drugs, albeit in the non-transplant setting.

Evidence suggests Vitamin D deficiency is correlated with poorer outcomes in this population; however, it is unknown if intensified Vitamin D supplementation improves outcomes. This clinical trial aims to address this question and will postulate the impact of Vitamin D on immunoregulatory functions and the hematopoietic niche microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age at time of registration to Step 1.
2. Patients must have history and physical exam within 28 days prior to registration.
3. Patients must have Zubrod/ECOG Performance Status ≤ 2.
4. Patients must have had a confirmed diagnosis of symptomatic MM (See Section 4.1) with measurable disease at the time of myeloma diagnosis that required systemic induction therapy prior to ASCT. Measurable disease is defined as measurable M protein in the serum (≥ 0.5g/dL) or urine (≥ 200 mg/24h) or serum free light chain assay (defined as ≥ 10 mg/dL [≥ 100 mg/L] on involved light chain) at the time of diagnosis. Patients with smoldering myeloma are not eligible until they have progressed to symptomatic myeloma.
5. Patients must be willing and able to take DVT prophylaxis (aspirin, low molecular weight heparin, warfarin, or equivalent oral anticoagulation) and comply with lenalidomide REMS program requirements.
6. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to registration. FCBP must agree to have a second pregnancy test within 24 hours prior to starting lenalidomide. Further, FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide. FCBP must also agree to ongoing pregnancy testing and must agree to not become pregnant for at least 3 months after the last dose of study treatment. A FCBP is a female who: 1) has achieved menarche (first menstrual cycle) at some point, 2) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).Men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy, during the study treatment and for 3 months after the last dose of study treatment.
7. Patients must have evidence of adequate renal function, as defined by (1) creatinine clearance (CrCl) ≥ 10 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula. Values must be obtained within 28 days prior to registration. Estimated creatinine clearance = (140 - age) x wt (kg) x 0.85 (if female) 72 x creatinine (mg/dl)
8. Patients must have adequate hepatic function defined by the following within 28 days prior to registration: Total bilirubin ≤ 1.5 x IULN (institutional upper limit of the norm) and AST and ALT ≤ 3.0 x IULN
9. Patients must be acceptable for transplant per institutional guidelines:
10. Patient's with human immunodeficiency virus (HIV) are eligible providing they are on effective antiretroviral therapy and have undetectable viral load at their most previous viral load test and within 6 months prior to registration.
11. Patients must be able to take and swallow oral medication (capsules) whole.
12. Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Any organ involvement by amyloidosis or evidence of amyloidosis related organ dysfunction.
2. Progressive disease at any time prior to registration.
3. Intolerance to the starting dose of lenalidomide (10 mg).
4. Prior allograft, prior organ transplant requiring immunosuppressive therapy, or have already received a previous autologous transplantation (e.g., requiring second ASCT at time of screening).
5. Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years.
6. Received any investigational agents within 14 days prior to registration.
7. Seropositive for Hepatitis B
8. Seropositive for Hepatitis C
9. Hypercalcemia (serum calcium level > 10.3 mg/dL) (institutional upper limit of the norm) at time of study entry.
10. Patients refractory to lenalidomide.
11. Patients that have received any investigational agents within 14 days prior to registration.
12. Any known impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). h known allergies to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To describe the lymphocyte subset analysis for the two treatment arms at 120 days post autologous stem cell transplant [120 days] | 120 days
  Evaluate absolute lymphocyte count and the difference in subset analysis (absolute CD4 count, absolute CD8 count) 120 days after ASCT

SECONDARY OUTCOMES:
3 year progression free survival | 3 years
  To report the 3-year progression-free survival for both treatment arms - maintenance Vitamin D vs. No maintnenace Vitamin D supplementation
Overall Response Rate post 120 days of ASCT | 120 Days
  report the overall response rate for both treatment arms 120 days after ASCT for adult patients with multiple myeloma.
Overall Response Rate after transplantation | Two Years
  To report the overall response rate for both treatment arms 2 years after transplantation
3 Year Overall Survival after transplantation | Three Years
  To report the 3-year overall survival for the two treatment arms after transplantation.
Minimal Residual Disease status | Randomization; 120 days after transplantation; two years after transplantation.
  To report the minimal residual disease status for the two treatment arms at randomization, and within 120 days after transplantation and 2 years after transplantation.
Vitamin D levels | Before autologous stem cell transplant; 120 days after transplantation; three years post-transplantation
  To report the vitamin D levels between the two treatments arms before autologous stem cell transplant, within 120 days, and 3-years post-transplantation
Adverse Event Reporting | Three years
  To describe the adverse events for the two treatment arms
Neutrophil and Platelet Engraftment and Transfusion Independence | After transplantation, an average of 30 days
  Time to neutrophil and platelet engraftment as well as transfusion independence after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Amany Keruakous, MD, Principal Investigator — Georgia Cancer Center at Augusta University
Locations (1):
- Georgia Cancer Center at Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No